CLINICAL TRIAL: NCT00006145
Title: A Phase III, Prospective, Randomized, Double-Blind Trial of Valganciclovir Pre-Emptive Therapy for Cytomegalovirus (CMV) Viremia as Detected by Plasma CMV DNA PCR Assay
Brief Title: Preventing Cytomegalovirus (CMV) Organ Damage With Valganciclovir in People With HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: A5030; 10170 (Registry Identifier: DAIDS ES); ACTG A5030; AACTG A5030
Record Dates: First submitted 2000-08-07; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Ganciclovir; Cytomegalovirus; Cytomegalovirus Infections; Administration, Oral; Antiviral Agents; Polymerase Chain Reaction; Viremia; DNA, Viral
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Viremia | interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
Cytomegalovirus (CMV) infection is a common opportunistic infection (OI) in HIV patients. The purpose of this study is to find out whether valganciclovir, an antiviral approved by the FDA for the treatment of CMV in the eye, is safe and effective in preventing CMV organ damage in people with HIV.

DETAILED DESCRIPTION:
CMV infection, most commonly of the retina (also known as CMV retinitis), is a common OI observed in HIV patients. Despite treatment, CMV retinitis can result in severe visual impairment and CMV disease is associated with reduced survival time. HIV patients receiving highly active antiretroviral therapy (HAART) for HIV infection who have CD4 counts less than 100 cells/mm3 may be at increased risk of CMV infection and its complications. Valganciclovir was approved by the FDA on March 29, 2001 for treatment of the symptoms of CMV retinitis in patients with weakened immune systems, including people with HIV and AIDS. This study will evaluate the safety and efficacy of valganciclovir in preventing CMV organ damage in HIV patients.

This study will last approximately 6 years. Step 1 is the longitudinal screening phase of the study. Patients at high risk for CMV disease who are enrolled in the study will be screened every 8 weeks for CMV in the blood; medical history assessment, physical examination, and blood work will occur at each visit. Additional blood collection to monitor HIV infection will occur every 16 weeks. Patients will undergo opthalmologic examination every 24 weeks. Patients who develop detectable CMV in their blood during Step 1 then enter Step 2 of the study.

In version 3.0 of this study, participants who test positive for CMV viremia or who are currently in Step 2 will be automatically enrolled into Step 4 and will be randomly assigned to one of two groups: 1) 900 mg valganciclovir twice daily for 3 weeks, followed by 900 mg valganciclovir daily, or 2) placebo. Participants will enter Step 3 if and when they develop CMV end-organ disease, at which point all participants will be offered 900 mg valganciclovir twice daily for 3 weeks, then 900 valganciclovir daily thereafter.

ELIGIBILITY:
Note: Per a recommendation from NIAID Therapeutic Trials Data Safety Monitoring Board (DSMB), this trial will close on 10/03/05. The DSMB has determined that the study will reach the primary objective. All participants not on valganciclovir must complete all study evaluations by 08/31/05; all participants taking valganciclovir must complete study evaluations by 10/03/05.

Inclusion Criteria for Step 1:

* HIV infected
* Viral load greater than 400 copies/ml
* CD4 count less than 100 cells/mm3
* Have taken HAART for 3 months or longer OR are not taking HAART and do not plan to start HAART for at least 3 months after study entry
* Have serum CMV IgG antibodies
* Have consent of parent or guardian if under 18 years of age
* Willing to use acceptable forms of contraception

Exclusion Criteria for Step 1:

* History of CMV end-organ disease
* Certain antiviral drugs for CMV prophylaxis within 8 weeks of study entry
* Pregnant or breastfeeding
* Currently require ongoing foscarnet or cidofovir. Limited courses of foscarnet or cidofovir for the treatment of diseases other than CMV are permitted if approved by the protocol chairs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350
Dates: Start 2000-08; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jacobson, MD, Study Chair — University of California, San Francisco and San Francisco General Hospital; David A. Wohl, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (57):
- United States (56):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Marin County Dept. of Health & Human Services, HIV/AIDS Program & Specialty Clinic, San Rafael, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Cornell CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Columbia Univ., HIV Prevention and Treatment Medical Ctr., New York, New York
  - AIDS Care CRS, Rochester, New York
  - McCree McCuller Wellness Ctr. at the Connection, Infectious Disease Unit, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Cleveland Clinic Foundation, Div. of Medicine, Infectious Diseases, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - Rhode Island Hosp., Providence, Rhode Island
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Univ. of Texas Southwestern Med. Ctr., Amelia Court Continuity Clinic, Dallas, Texas
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Cocohoba JM, McNicholl IR. Valganciclovir: an advance in cytomegalovirus therapeutics. Ann Pharmacother. 2002 Jun;36(6):1075-9. doi: 10.1345/aph.1A393. PMID 12022911
- [Background] De Clercq E. Antiviral drugs in current clinical use. J Clin Virol. 2004 Jun;30(2):115-33. doi: 10.1016/j.jcv.2004.02.009. PMID 15125867
- [Background] Erice A, Tierney C, Hirsch M, Caliendo AM, Weinberg A, Kendall MA, Polsky B; AIDS Clinical Trials Group Protocol 360 Study Team. Cytomegalovirus (CMV) and human immunodeficiency virus (HIV) burden, CMV end-organ disease, and survival in subjects with advanced HIV infection (AIDS Clinical Trials Group Protocol 360). Clin Infect Dis. 2003 Aug 15;37(4):567-78. doi: 10.1086/375843. Epub 2003 Jul 29. PMID 12905142
- [Background] Reusser P. Oral valganciclovir: a new option for treatment of cytomegalovirus infection and disease in immunocompromised hosts. Expert Opin Investig Drugs. 2001 Sep;10(9):1745-53. doi: 10.1517/13543784.10.9.1745. PMID 11772283
- [Result] Wohl DA, Kendall MA, Andersen J, Crumpacker C, Spector SA, Feinberg J, Alston-Smith B, Owens S, Chafey S, Marco M, Maxwell S, Lurain N, Jabs D, Benson C, Keiser P, Jacobson MA; A5030 Study Team. Low rate of CMV end-organ disease in HIV-infected patients despite low CD4+ cell counts and CMV viremia: results of ACTG protocol A5030. HIV Clin Trials. 2009 May-Jun;10(3):143-52. doi: 10.1310/hct1003-143. PMID 19632953